CLINICAL TRIAL: NCT01216475
Title: Comparison of Small Incision Lenticule Extraction (SMILE) and VisuMax Femtosecond Laser In Situ Keratomileusis (FemtoLASIK): A Randomized, Non-inferiority Trial
Brief Title: Randomized, Non-inferiority Trial Comparing SMILE and LASIK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Federico Luengo Gimeno, Prof Jod Mehta, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R788/72/2010
Record Dates: First submitted 2010-09-08; First posted 2010-10-07 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Myopia; Astigmatism; Hypermetropia
MeSH Terms: conditions — Myopia; Astigmatism; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femtosecond LASIK (Active Comparator): 2 lasers refractive procedure
  Interventions: Procedure: Femtosecond LASIK
- SMILE (Experimental): Small incision lenticule extraction (SMILE)
  Interventions: Procedure: Small incision lenticule extraction (SMILE)

INTERVENTIONS:
Procedure: Femtosecond LASIK — LASIK consists of two steps: the first step involves the formation of a corneal flap and the second one is when the excimer ablation is performed in the corneal stromal bed. Femtosecond lasers (FL) have been widely used in LASIK surgery to fashion the corneal flap. The laser will cut a lamellar followed by a vertical corneal incision. We are able to produce a vertical cut since the Femtosecond laser can deliver laser pulses of 1 micron diameter at a preselected depth in the cornea, which then expands to 2 to 3 microns with the formation of a cavitation bubble. These pulses create micro-photodisruption of the corneal tissue by the formation of an expanding bubble of carbon dioxide and water, which in turn cleaves the tissue and creates a plane of separation. The flap is then removed to expose the stroma and the refractive treatment is done by the excimer laser over the denuded stroma.
  Other Names: Blade-less LASIK
  Arms: Femtosecond LASIK
Procedure: Small incision lenticule extraction (SMILE) — Patient's eye will be centered and docked with the curved interface cone before application of suction fixation. First, the posterior surface of the refractive lenticule (spiral in), then the lenticule border is created. The anterior surface of the refractive lenticule (spiral out) is then formed which extended beyond the posterior lenticule diameter by 0.5mm to form the anterior flap and is followed by a rim cut. After the suction is released, a Siebel spatula is inserted under the flap near the hinge before the flap is seperated and reflected. The edge of the refractive lenticule is separated from the stromal bed with a sinsky hook and the posterior border of the lenticule gently separated with the Siebel spatula and removed through small incision.
  Arms: SMILE

SUMMARY:
Background: Small Incision Lenticule Extraction or SMILE is a novel form of 'flapless' corneal refractive surgery that was adapted from Refractive Lenticule Extraction (ReLEx). SMILE uses only one femtosecond laser to complete the refractive surgery, potentially reducing surgical time, side effects and cost. If successful, SMILE could potentially replace the current, widely practiced Laser In-situ Keratomileusis or LASIK. The aim of this study is to evaluate whether SMILE is non-inferior to LASIK in terms of refractive outcomes at 3-months post-operatively.

Methods/ Design: Single tertiary center, parallel group, single-blinded, paired-eye design, non-inferiority, randomized controlled trial. Participants who are eligible for LASIK will be enrolled for study after informed consent. Each participant will be randomized to receive SMILE and LASIK in each eye. Our primary hypothesis (stated as null) in this non-inferiority trial would be that SMILE differs from LASIK in adults (>21 years old) with myopia (> -3.00D) at a tertiary eye center in terms of refractive predictability at 3 months post-operatively. Our secondary hypothesis (stated as null) in this non-inferiority trial would be that SMILE differs from LASIK in adults (>21 years old) with myopia (> -3.00D) at a tertiary eye center in terms of other refractive outcomes (efficacy, safety, higher-order aberrations) at 3 months post-operatively. Our primary outcome is refractive predictability, which is one of several standard refractive outcomes, defined as the proportion of eyes achieving a postoperative spherical equivalent (SE) within ±0.50 diopter (D) of the intended target. Randomization will be performed using random allocation sequence generated by a computer with no blocks or restrictions, and implemented by concealing the number-coded surgery within sealed envelopes until just before the procedure. In this single-blinded trial, subjects and their caregivers will be blinded to the assigned treatment in each eye.

Discussion: This novel trial will provide information on whether SMILE has comparable, if not superior, refractive outcomes compared to the established LASIK for myopia, thus providing evidence for translation into clinical practice.

DETAILED DESCRIPTION:
Surgical correction for refractive errors may be performed by a number of procedures. Laser correction involves procedures such as EpiLASIK, LASIK or conductive keratoplasty, while lens based corrections involve the use of phakic intra-ocular lenses. Despite the emergence of other procedures, due to its fast visual rehabilitation and painless postoperative course, LASIK is still the procedure of choice for both patients and refractive surgeons.

LASIK consists of two steps: the first step involves the formation of a corneal flap and the second one is when the excimer ablation is performed in the corneal stromal bed. Femtosecond lasers (FL) have been widely used in LASIK surgery to fashion the corneal flap. The laser will cut a lamellar followed by a vertical corneal incision. We are able to produce a vertical cut since the Femtosecond laser can deliver laser pulses of 1 micron diameter at a preselected depth in the cornea, which then expands to 2 to 3 microns with the formation of a cavitation bubble. These pulses create micro-photodisruption of the corneal tissue by the formation of an expanding bubble of carbon dioxide and water, which in turn cleaves the tissue and creates a plane of separation. The flap is then removed to expose the stroma and the refractive treatment is done by the excimer laser over the denuded stroma. The advantages of femtosecond laser over microkeratome LASIK flaps have been reduced postoperative dry eye symptoms, less chance of dislocation from trauma and reduced incidence of button holes or free caps.

Even though femto-LASIK has demonstrated good efficacy, it can still be asssociated with side effects found in standard LASIK e.g. glare, haloes, dry eye and still requires the use of two laser machines, one for the flap the other for the excimer ablation. This increases the length of time of the overall procedure and the costs.

Recently, a new "one laser" refractive surgery has been proposed: Femtosecond Lenticule Ex-traction (FLEx). It consists of performing the entire refractive procedure without an excimer laser. The Femtosecond laser creates four stromal incisions to create a corneal lenticule and a corneal flap. The size and shape of the lenticule is calculated based on the patient refractive error. The lenticule is separated from the flap above and the rest of the cornea below using a small spatula. Following this, the lenticule is grasped with a forceps and extracted from the eye. Finally, the flap is repositioned and the interface washed. At this time the refractive error is already corrected without the use of a second laser.

The advantages of FLEx treatment are shortened length of the refractive procedure, reduced patient inconvenience from moving from one laser to another, reduced risk of intraoperative infections and more accurate ablation since the patient need to fixate only once.

Currently there are no publications comparing FLEx to LASIK, hence this study will be unique in the fact that the paired eye approach will act as an internal patient control to assess the objective and subjective outcomes in patients following both these procedures.

The study will be a prospective randomized trial of patients comparing SMILE (a variation of FLEx) with LASIK to treat their myopic refractive error. One eye will be randomized for SMILE and other eye for LASIK. Each procedure will be performed sequentially. Randomization will be performed by a random number generator, and assignment concealed in envelopes.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older.
2. Cycloplegic spherical equivalent of >-2.00D
3. Refractive cylinder -4.00 D or less, Anisometropia of >1D
4. Best spectacle corrected visual acuity (BSCVA) of 6/12 or better in BOTH eyes.
5. Spherical or cylindrical error has progressed at -0.50D or less per year from date of baseline measurement.
6. Contact lens wearers must have removed contact lenses at least two (2) weeks before the baseline measurement.
7. No evidence of irregular astigmatism on corneal topography.
8. Available to attend post-operative examinations for a 3 month period.

Exclusion Criteria:

1. Progressive or unstable myopia and/or astigmatism.
2. Clinical or corneal topographic evidence of keratoconus.
3. Residual, recurrent or active ocular disease such as uveitis, severe dry eyes, severe allergic eye disease, glaucoma, visually significant cataract and retinal disease.
4. Previous corneal surgery or trauma within the corneal flap zone.
5. Patent corneal vascularization within 1mm of the corneal flap zone.
6. Taking systemic medications likely to affect wound healing, such as corticosteroids and antimetabolites.
7. Systemically immunocompromised.
8. Systemic disease likely to affect wound healing, such as diabetes, connective tissue disease and severe atopy.
9. Pregnant or nursing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Refractive predictability | 3 months Post-operative
  Defined as the proportion number of eyes achieving a postoperative spherical equivalent (SE) within ±0.50 diopter (D) of the intended target.

SECONDARY OUTCOMES:
Efficacy | 3 months Post-operative
  Defined as the proportion number of eyes achieving a unaided visual acuity (UAVA) of 20/20 or better postoperatively
Safety | 3 months Post-operative
  Defined as the proportion number of eyes that lost or gained 1 or more lines of postoperative best-corrected visual acuity (BCVA) relative to the preoperative BCVA
Contrast sensitivity | 3 months Post-operative
  Tested using the Vision Contrast Test System (VCTS) chart (VCTS 6500 contrast sensitivity Chart) in 6 spatial frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Donald T Tan, FRCS(Ed),, Study Director — Singapore National Eye Centre; Jodhbir S Mehta, FRCS (ed), Principal Investigator — SNEC
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sekundo W, Kunert K, Russmann C, Gille A, Bissmann W, Stobrawa G, Sticker M, Bischoff M, Blum M. First efficacy and safety study of femtosecond lenticule extraction for the correction of myopia: six-month results. J Cataract Refract Surg. 2008 Sep;34(9):1513-20. doi: 10.1016/j.jcrs.2008.05.033. PMID 18721712
- [Derived] Ang M, Tan D, Mehta JS. Small incision lenticule extraction (SMILE) versus laser in-situ keratomileusis (LASIK): study protocol for a randomized, non-inferiority trial. Trials. 2012 May 31;13:75. doi: 10.1186/1745-6215-13-75. PMID 22647480